CLINICAL TRIAL: NCT02895984
Title: Reducing Hazardous Alcohol Use in Social Networks Using Targeted Intervention
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: Oregon Research Institute (Other); Smith College (Other); University of Massachusetts, Worcester (Other)
Responsible Party: Principal Investigator, Nancy Barnett, Principal Investigator, Brown University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1R01AA02352201A1
Record Dates: First submitted 2016-08-22; First posted 2016-09-12 (Estimated); Last update posted 2019-08-02 (Actual); Status verified 2019-07

CONDITIONS: Alcohol Consumption; Alcohol Abuse
Keywords: Social network analysis; Brief Motivational Interviewing; College Students
MeSH Terms: conditions — Alcohol Drinking; Alcoholism | interventions — Ethanol; Methods; Body Mass Index

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Brief Motivational Intervention (BMI) (Experimental): The intervention recipients in the BMI group will receive a 1-hour single-session alcohol intervention (BMI) with personalized normative feedback.
  Interventions: Behavioral: Single-session alcohol intervention (BMI)
- Natural History Control (NHC) (No Intervention): Students in the NHC group will receive no contact.

INTERVENTIONS:
Behavioral: Single-session alcohol intervention (BMI) — The intervention recipients will receive a 1-hour individual BMI. The BMI will follow the central principles of Motivational Interviewing (MI) and will include all the components determined to be efficacious in existing multi-component BMIs (e.g., personalized feedback on indicators of alcohol-related risk, including signs of alcohol dependence and family history of alcohol risk; normative comparisons of the participant's alcohol consumption with same-sex peers in his/her dorm and throughout campus, and protective behavioral strategies). Additional components will include reviewing the pros and cons of the participant's current pattern of alcohol use, providing estimates of the participant's recent Blood Alcohol Concentration (BAC), and providing information about risks of specific negative outcomes at different levels of drinking. Participants will identify goals for behavior change, and with the counselor will develop a plan to achieve the goals and to address barriers to success.
  Arms: Brief Motivational Intervention (BMI)

SUMMARY:
Alcohol use is almost ubiquitous on college campuses and first-year students are at particularly high risk of alcohol-related harm when they first make the transition to college. Peers are important agents in socializing both healthy and unhealthy behaviors, but despite the clear role of peer behavior in the maintenance of college problem drinking, there have been no efforts to measure the effect of individual change on the reduction of alcohol-related risks in the broader student body. That is, despite the importance of social connections for inducing and maintaining alcohol use in youth, intervention approaches have not measured nor capitalized on the potential of social influences for changing this problem behavior. It is essential that we understand the indirect effects of individual interventions and the impact such interventions have on the social structure and social connections. The best way to evaluate such effects is to use a research design that experimentally manipulates drinking using the best available intervention and measures its effects on the social network and its members.

The purpose of this research is to investigate whether using an established individual Brief Motivational Intervention (BMI) administered to a small number of influential network members embedded in a social network significantly reduces heavy drinking and alcohol consequences among close peers who do not receive any intervention. In addition, the investigators will investigate social influence mechanisms of this transmitted effect, investigate how specific types of network connections and relationships moderate the indirect intervention effect, and investigate the effects of the intervention on network position and structure. First-year students at Brown will be enrolled and assessed early in their fall 2016 academic semester. Heavy drinkers in each dormitory who are in the top quartile of betweenness centrality, a social network construct that reflects high connectivity and potential influence, will either receive BMI or serve as controls, according to their dormitory's intervention assignment. All participants will be assessed again 5 and 12 months after baseline to measure changes in behavior and in peer ties. The long-term objective of this research is to understand how peer influences function in social networks in order to leverage those mechanisms to reduce problematic alcohol use in heavy drinking populations.

DETAILED DESCRIPTION:
The proposed design and network analytic methods will allow the investigators to investigate the extent to which an intervention conducted with careful attention to network connection is transmitted to others (Aim 1), how those effects occur (Aim 2), conditions under which those effects are more likely (Aim 3), and how the connections themselves change as a function of the intervention (Aim 4).

AIM 1. To investigate the efficacy of targeted Brief Motivational Intervention for reducing heavy drinking and alcohol consequences in network members who received no intervention. The investigators expect that heavy drinking participants residing in dormitories assigned to BMI but who receive no intervention will show lower frequency of heavy drinking and alcohol consequences at follow-up than their comparison group in NHC dormitories (n = 480; 240 in each condition).

AIM 2. To identify the social influence mechanisms through which the intervention effect is conveyed. The investigators expect that reductions in the following social influence mechanisms will mediate the indirect intervention effect: (1) behavioral modeling of heavy drinking; (2) social reinforcement for drinking or not drinking; (3) offers and provision of alcohol; (4) the perception of peer heavy drinking (descriptive norms); and (5) the perception of peer approval of heavy drinking (injunctive norms).

AIM 3. To identify the network and relationship features that moderate intervention efficacy.

3A. Proximity to Intervention. The investigators expect that heavy drinking network members who: (1) have first-degree ties (i.e., a direct tie) with intervention recipients, (2) have a higher proportion of intervention recipients in their close network (i.e., have the highest exposure to transmitted intervention effects), and (3) have an intervention recipient as a roommate will show the strongest indirect intervention effect.

3B. Quality of Peer Relationships. The investigators expect that stronger relationships with intervention recipients as measured by: (1) best-friend status, (2) higher perceived relationship closeness, (3) higher perceived social support, and (4) reciprocated network nominations, will be related to greater indirect intervention effects.

AIM 4. To investigate the intervention effect on personal-level network position and on drinking-based selection in the network.

4A. Network position. Differences between the intervention recipients in the BMI and NHC groups at follow-up will be investigated on: (1) betweenness centrality (how often the participant falls on the shortest path between two others) and (2) prestige (number of nominations of the participant by others). There is little literature on how network positions change following behavioral intervention, so directional hypotheses are not proposed.

4B. Drinking-based selection. At follow-up, the investigators expect less drinking-based selection in the BMI group compared to the NHC group.

ELIGIBILITY:
Inclusion Criteria:

* Students enrolled as full-time first-year students at Brown University

Exclusion Criteria:

* Students not enrolled as full-time first-year students at Brown University

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1424 (Actual)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-10-31 (Actual); Study Completion 2017-10-31 (Actual)

PRIMARY OUTCOMES:
Change in frequency of heavy drinking | baseline, 5-months post baseline, 12-months post-baseline
  Heavy episodic drinking (HED) frequency is defined as the number of occasions in which participants drank 4+ (for females) or 5+ (for males) standard alcoholic drinks per drinking occasion during the past 30 days.
Change in endorsed negative alcohol consequences | baseline, 5-months post baseline, 12-months post-baseline
  24-item (no/yes) response on the Brief Young Adult Alcohol Consequences Questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Nancy P Barnett, PhD, Principal Investigator — Brown University

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ott MQ, Clark MA, Balestrieri SG, Gamarel KE, Barnett NP. Social Networks and Sexual and Gender Minority Disparities in Alcohol Use and Consequences Among First-Year College Students. LGBT Health. 2022 Oct;9(7):489-495. doi: 10.1089/lgbt.2019.0225. Epub 2022 Jun 21. PMID 35727117
- [Derived] Barnett NP, Clark MA, Kenney SR, DiGuiseppi G, Meisel MK, Balestrieri S, Ott MQ, Light J. Enrollment and assessment of a first-year college class social network for a controlled trial of the indirect effect of a brief motivational intervention. Contemp Clin Trials. 2019 Jan;76:16-23. doi: 10.1016/j.cct.2018.10.015. Epub 2018 Nov 1. PMID 30391343
- [Derived] DiGuiseppi GT, Meisel MK, Balestrieri SG, Ott MQ, Clark MA, Barnett NP. Relationships between social network characteristics, alcohol use, and alcohol-related consequences in a large network of first-year college students: How do peer drinking norms fit in? Psychol Addict Behav. 2018 Dec;32(8):914-921. doi: 10.1037/adb0000402. Epub 2018 Sep 27. PMID 30265059
- [Derived] Kenney SR, DiGuiseppi GT, Meisel MK, Balestrieri SG, Barnett NP. Poor mental health, peer drinking norms, and alcohol risk in a social network of first-year college students. Addict Behav. 2018 Sep;84:151-159. doi: 10.1016/j.addbeh.2018.04.012. Epub 2018 Apr 16. PMID 29684764